CLINICAL TRIAL: NCT00580528
Title: Modifying Lifestyle in Prehypertensive Older Rural Women
Brief Title: Reducing Blood Pressure in Prehypertensive Older Rural Women Also Known as Wellness for Women: DASHing Toward Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0352-05-FB; 5R01NR004861-06 (NIH); 31-4334-0124 (Other Grant/Funding Number: National Institute of Nursing Research)
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pre-Hypertension
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Tailored internet newsletters (Experimental): Tailored newsletters delivered via the Internet with content for improving eating and activity to reduce blood pressure.
  Interventions: Behavioral: Tailored Internet Newsletters
- 2 Tailored print newsletters (Experimental): Tailored print newsletters delivered via the mail with content for improving eating and activity to reduce blood pressure.
  Interventions: Behavioral: Tailored print newsletters delivered via mail
- 3 No newsletters (No Intervention): Participants receive no newsletters

INTERVENTIONS:
Behavioral: Tailored Internet Newsletters — Tailored newsletters delivered via the Internet with content for improving eating and activity to reduce blood pressure
  Arms: 1 Tailored internet newsletters
Behavioral: Tailored print newsletters delivered via mail — Tailored Newsletters with content to improve eating and activity to reduce blood pressure
  Arms: 2 Tailored print newsletters

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a theory-based intervention tailored to constructs in the Health Promotion Model and delivered by two distance modes to achieve improvement in healthy eating and physical activity for the control of blood pressure (BP) among an underserved and vulnerable population of prehypertensive rural women aged 50 to 69.

DETAILED DESCRIPTION:
Hypertension (HTN), a major health problem in the US, is the most prevalent modifiable risk factor for cardio-vascular disease (CVD), the leading killer of women. The incidence of HTN in women increases markedly after menopause, equaling or exceeding that in men. The prehypertension category of blood pressure (BP) -- systolic BP of 120-139 mm Hg or diastolic BP of 80-89 mm Hg -- designates individuals at high risk of developing HTN. Prehypertensive women are not candidates for drug therapy, but for lifestyle modifications to prevent progression to HTN and CVD. Recommended lifestyle modifications include adoption of the Dietary Approaches to Stop Hypertension (DASH) diet that is high in fruits, vegetables and low fat dairy products; dietary sodium reduction; regular endurance physical activity supplemented by resistance exercise; and weight reduction by those who are overweight or obese. A few studies of face-to-face individual and/or group interventions have demonstrated that these lifestyle modifications could lower BP over 6 months in pre-hypertensive individuals. There remains a need to develop distance delivery methods to target rural women with similar behavioral interventions to lower BP. This competitive renewal application will build upon our current work in which we demonstrated that computer-generated print (mailed) newsletters tailored to constructs in the Health Promotion Model (HPM) resulted in significant and clinically important changes in behavioral and biomarkers of healthy eating and physical activity in a general population of rural midlife/older women. The proposed randomized controlled trial will evaluate Internet versus mailed print delivery methods for delivering theory-based tailored newsletters to encourage lifestyle change for BP reduction. A sample of 275 prehypertensive rural women aged 50-69 will be randomly assigned 2:2:1 to receive a) tailored messages delivered via the Internet and brief telephone counseling, b) tailored print newsletters delivered via mail and brief telephone counseling, or c) initial standard advice only. Results of this study may lead to expanded access to lifestyle guidance via the Internet by other populations.

ELIGIBILITY:
Inclusion Criteria:

* women aged 50-69
* BP in prehypertensive range (SBP 120-139 or DBP 80-89 mm Hg)
* speak and read English (including ESL)
* able to communicate over the telephone
* able to use a computer with minimal assistance
* have access to the Internet
* have access to a VCR or DVD player
* able to walk without an assistive device
* answer 'no' to all questions on the Physical Activity Readiness Questionnaire (PAR-Q) or obtain clearance from their physician

Exclusion Criteria:

* in the maintenance stage of readiness for change in both components of physical activity and all three components of healthy eating behaviors
* more than 14 alcoholic drinks per week
* taking anti-hypertensive medication, including diuretics
* taking cortisone
* currently enrolled in a formal program of cardiac rehabilitation or undergoing physical rehabilitation
* unable to walk one mile continuously without stopping to rest
* current cancer treatment
* other physical or medical restrictions that would preclude following the JNC7 recommendations for moderate physical activity and healthy eating.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2011-05-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 24 months
  Blood pressure with the criterion of normotensive status

SECONDARY OUTCOMES:
Daily moderate physical activity and strength enhancing/maintenance activities | 24 months
  Engaging regularly, preferably daily, in sustained or intermittent (10 minute bouts) moderate physical activity for at least 30 minutes per day and performing physical activities that enhance and maintain muscular strength at least twice a week.
DASH diet goals | 24 months
  Meeting the DASH diet's average daily goals of no more than 27% of calories from fat, less than 7% of calories from saturated fat 4-5 servings of fruits, 4-5 servings of vegetables, 2-3 servings of low fat dairy products and no more than 2400 mg. sodium.

CONTACTS AND LOCATIONS:
Overall Officials: Carol H Pullen, EdD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Hageman PA, Pullen CH, Hertzog M, Boeckner LS. Effectiveness of tailored lifestyle interventions, using web-based and print-mail, for reducing blood pressure among rural women with prehypertension: main results of the Wellness for Women: DASHing towards Health clinical trial. Int J Behav Nutr Phys Act. 2014 Dec 6;11:148. doi: 10.1186/s12966-014-0148-2. PMID 25480461
- [Derived] Hageman PA, Pullen CH, Hertzog M, Boeckner LS, Walker SN. Associations of cardiorespiratory fitness and fatness with metabolic syndrome in rural women with prehypertension. J Obes. 2012;2012:618728. doi: 10.1155/2012/618728. Epub 2012 Nov 25. PMID 23227315